CLINICAL TRIAL: NCT03921320
Title: Evaluation of Compensatory Sweating After Unilateral Videothoracoscopic Sympathectomy of the Dominant Side or Sequential Bilateral Videothoracoscopic Sympathectomy: a Multicentric Randomized Trial
Brief Title: Compensatory Sweating After Unilateral Sympathectomy on the Dominant Side or Bilateral Sequential Sympathectomy
Acronym: Universusbi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Miguel L. Tedde, Thoracic surgeon, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Usaopaulo04032019
Record Dates: First submitted 2019-03-11; First posted 2019-04-19 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Hyperhidrosis Primary Focal Palms
Keywords: Hyperhidrosis; Sympathectomy; Sweating
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to be submitted to sequential bilateral sympathectomy or unilateral sympathectomy on the dominant side. After 4 to 6 months participants of the unilateral group can make the contralateral sympathectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bilateral sympathectomy (Active Comparator): Bilateral sequential (one surgical procedure) videothoracoscopic R4 sympathectomy
  Interventions: Procedure: Bilateral sequential sympathectomy
- Unilateral sympathectomy (Experimental): Unilateral videothoracoscopic R4 sympathectomy on the right (dominant) side
  Interventions: Procedure: Unilateral sympathectomy
- Contralateral sympathectomy (Experimental): Unilateral videothoracoscopic R4 sympathectomy on the left (contralateral) side
  Interventions: Procedure: Contralateral sympathectomy

INTERVENTIONS:
Procedure: Bilateral sequential sympathectomy — Bilateral videothoracoscopic sequential R4 sympathectomy
  Arms: Bilateral sympathectomy
Procedure: Unilateral sympathectomy — Unilateral videothoracoscopic R4 sympathectomy in dominant side (right side)
  Arms: Unilateral sympathectomy
Procedure: Contralateral sympathectomy — Contralateral (left side) videothoracoscopic R4 sympathectomy
  Arms: Contralateral sympathectomy

SUMMARY:
The standard treatment for palmar hyperhidrosis is bilateral sequential thoracic sympathectomy. High rates of compensatory sweating due to the surgical procedure are described in the literature. In the search for a reduction in this side effect, it is possible that unilateral sympathectomy in the dominant side obtains acceptable results and leads to less compensatory sweating with improvement of the quality of life. The aim of this study it to compare the intensity of compensatory sweating due to the standard treatment, that is, bilateral sequential videothoracoscopic sympathectomy in relation to unilateral thoracic sympathectomy on the dominant side.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index equal to or less than 28;
* Exclusive palmar hyperhidrosis or palmar hyperhidrosis associated with axillary and / or plantar hyperhidrosis;

Exclusion Criteria:

* Being sinister (or left-handed);
* Craneo-f acial or generalized hyperhidrosis;
* Coagulopathies;
* Previous thoracic surgery;
* Other comorbidities such as cardiological, metabolic, infectious or neoplastic diseases;
* Pregnancy;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change of sweating intensity | Change from baseline sweating to 6 months after surgery
  To utilize the HDSS questionnaire to assessment of sweating intensity change in patients with palmar hyperhidrosis treated by bilateral sequential thoracic sympathectomy

SECONDARY OUTCOMES:
Change of sweating intensity | Change from baseline sweating to 6 months after sympathectomy
  To utilize the HDSS questionnaire to assessment of sweating intensity change in patients with palmar hyperhidrosis submitted to unilateral sympathectomy on the dominant (right) side
Change of sweating intensity | Change from baseline sweating to 6 months after surgery
  To utilize the HDSS questionnaire to assessment of sweating intensity change in patients submitted to contralateral (left side) sympathectomy after unilateral sympathectomy on the dominant side

OTHER OUTCOMES:
Change of Quality of life | Change from baseline quality of life to 6 months after surgery
  To utilize the HidroQOL questionnaire to evaluate the change in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Miguel L Tedde, MD, PhD, Study Chair — Thoracic Surgeon, InCor, FMUSP
Locations (10):
- Brazil (10):
  - Hospital Universitário da Universidade Federal do Amazonas, Manaus, Amazonas
  - Hospital Geral Dr. Cesar Cals, Fortaleza, Ceará
  - Hospital Santa Isabel, Salvador, Estado de Bahia
  - Instituto Hospital de Base, Brasília, Federal District
  - Hospital Julia Kubitschek, Belo Horizonte, Minas Gerais
  - Hospital Maternidade Terezinha de Jesus, Juiz de Fora, Minas Gerais
  - Hospital Universitário Oswaldo Cruz, Recife, Pernambuco
  - Hospital Universitário Pedro Ernesto, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Onofre Lopes, Natal, Rio Grande do Norte
  - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Grande do Sul